CLINICAL TRIAL: NCT03670511
Title: Validation and Predictive Equation for Sit-to-stand Test in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, G.Reychler, Physiotherapist, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STSTvalid
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sit-to-stand (Experimental)
  Interventions: Other: sit-to-stand test
- six minute walking test (Active Comparator)
  Interventions: Other: six minute walking test

INTERVENTIONS:
Other: sit-to-stand test — to sit and stand from a chair
  Arms: sit-to-stand
Other: six minute walking test — to walk for six minutes
  Arms: six minute walking test

SUMMARY:
Validation and development of predictive values for the one minute sit-to-stand test in children between 6 and 18 years.

ELIGIBILITY:
Inclusion Criteria:

* participation in the national physical education program at school
* free of physical activity during one hour preceding the experiments

Exclusion Criteria:

* diagnosis of chronic lung, cardiac or neuromuscular disease
* BMI higher than 85th percentile for children of the same age and sex
* a motor disability based on parents' answer to standardized questions.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 397 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
number of sit-to-stand | 1 minute

SECONDARY OUTCOMES:
pulsed oxygen saturation | 1 minute
heart rate | 1 minute

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No